CLINICAL TRIAL: NCT03118271
Title: Comparison of the Effect of Lumbar Traction, Spinal Manipulation, and Surgery in the Treatment of Lumbar Disc Herniation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Two authors changed their jobs.
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20160806R
Record Dates: First submitted 2017-04-07; First posted 2017-04-18 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2018-04

CONDITIONS: Lumbar Disc Herniation; Lumbar Traction; Spinal Manipulation; Lumbar Surgery
Keywords: lumbar disc herniation; lumbar traction; spinal manipulation; lumbar surgery
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Manipulation, Spinal; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- lumbar traction (Active Comparator): Treatment with lumbar traction is via an OPD base. It comprised a 20 min. treatment session over a period of 2 months. If the symptoms subside before the end of 2 months' treatment, lumbar traction will be discontinued, and the treatment duration and number of treatment session will be recorded. The frequency of treatment is 3 times per week. Treatment method is according to the common clinical guidelines, starting from 25% of the subject's body weight and steadily increasing to 50% of body weight. Before traction, heat therapy will be applied to the low back of the subject, and electric therapy will also be given to the painful areas. The treatment will be conducted by the same physiotherapist.
  Interventions: Device: lumbar traction
- spinal manipulation (Active Comparator): Spinal manipulation will be performed by a spinal manipulator (Dr. Tso-Liang Wang) who was graduated from Los Angeles College of Chiropractic. Before performing spinal manipulation, he will exam the patient's whole body throughly, especially focusing on the lumbo-pelvic-hip region. What he exams includes pelvic and spinal alignment, tension of soft tissues, tissue texture, joint mobility, movement patterns, and muscle power. The manipulation is started with release of the hypertonic myofascial structures and thus normalize the myofascial tension of the lumbo-pelvic-hip region. Then he will align the lumbar spine, pelvis and hip joint three-dimensionally according to the findings of his examination on the same day. The manipulation will be performed up to 8 times within one month (no more than 2 manipulations a week). If the symptoms subside before the end of one-month' treatment, the manipulation is discontinued and the number of treatment session will be recorded.
  Interventions: Procedure: spinal manipulation
- surgery (Active Comparator): General anesthesia, the patient will be put in the prone and abdomen-free position. A 4-cm midline longitudinal incision will be made over the spinous processes of the L3-5 levels. It will be deepened through the fat and fascia in line with the skin incision to reach the spinous processes.The paraspinous muscles will be dissected subperiosteally down the spinous processes and along the lamina to the facet joints. Laminectomy will be done carefully at the herniated disc level for posterior decompression. The ligamentum flavum will be excised to expose the dural sac.Using blunt dissection, the investigators carefully continue down the lateral side of the dura to the floor of the spinal canal; the investigators retract the dura and its nerve root medially. After the posterior aspect of the disc space is revealed, the affected disc will be removed and discotomy will be performed.The wound will be closed in the routine fashion after meticulous hemostasis and normal saline irrigation.
  Interventions: Procedure: surgery

INTERVENTIONS:
Device: lumbar traction
  Arms: lumbar traction
Procedure: spinal manipulation
  Arms: spinal manipulation
Procedure: surgery
  Arms: surgery

SUMMARY:
To compare the effect of lumbar traction, lumbar spinal manipulation and lumbar surgery in the treatment of LDH.

DETAILED DESCRIPTION:
Back pain is the second leading cause of work absenteeism (after upper respiratory tract complaints) and results in more lost productivity than any other medical condition. The lifetime prevalence of back pain exceeds 70% in most industrialized countries,and the 1-year prevalence for an episode of acute low back pain (LBP) has been estimated to be 65%. Sciatica is present in about 25% of those with LBP, and one of the major cause of sciatica is herniation of intervertebral disc (HIVD) of the lumbosacral spine or lumbar disc herniation (LDH). In the United Kindom, the estimated prevalence of LDH is from 1% to 3%. Although 95% of LBP patients recovered in 12 weeks, recurrent pain and disability were common and occurred in 12% over the 18-month observation period.

Disc herniation may be purely annular, purely nuclear, or consist of a combination of annular and nuclear tissues. Nuclear disc herniation track posteriorly between the anterior surface of the posterior longitudinal ligament and the posterior surfaces of the annulus and vertebral body and then into the spinal canal. Disc herniation may be described as protrusion or extrusion (or sequestration, if the displaced disc material has lost completely any continuity with the parent disc); contained or uncontained.

The usual presenting complaint is acute or chronic intermittent LBP with or without sciatica, which is radiating pain in a dermatomal distribution and classically described as a burning, stabbing, or electric sensation, sometimes accompanied with paresthesia. Central disc herniations or herniation that have migrated can each result in a mixed clinical picture or, alternately, signs of stenosis may predominate. The mechanism of pain is mutifactorial, involving mechanical stimulation of the nerve endings in the outer annulus, direct compression on the posterior longitudinal ligament, dura, or nerve root, and/or the chemical inflammatory cascade induced by the exposed nucleus pulposus or annulus fibrosis.The classic straight leg raising (SLR) test or Lasegue test is thought to be a useful clinical test to demonstrate an inflammatory compressive process across single or multiple spinal nerve roots.

Magnetic resonance imaging (MRI) has become the examination of choice for diagnosing LDHs.It has the advantage of having no known side effects or morbidity, no radiation exposure, and is noninvasive. The sensitivity and specificity of MRI in detecting annular tears, disc herniation, and nerve root swelling has been confirmed in several studies. MRI findings have been correlated to clinical findings and are strong predictors of surgical outcomes. However, morphological abnormalities demonstrated by MRI do not always reflect LBP or sciatica. MRI should be interpreted with consideration of full clinical signs, symptoms, and other relevant background.

Treatment of LDH consists of operative and non-operative treatments. Non-operative care of LDH includes a wide range of different methods: lumbar supports, bed rest, oral analgesics and muscle relaxants, lumbar traction, therapeutic exercise, spinal manipulation, epidural steroid injections, and behavioral therapy.

Lumbar traction is a very popular therapy for treatment of LDH in our country. Patients would be placed in traction with the expectation that stretching of the lumbar area would result in distraction and elongation of the structural elements and resolution of pain. Other physiological effects of lumbar traction including decrease in the intra-disc pressure, relief of muscle spasm , reduction of prolapsed disc and forcing patients to bed rest. Despite favorable outcomes have been reported previously,there are few scientifically rigorous studies in the literature that allow the effect of traction to be distinguished from the natural history of the pathology being treated.

Spinal manipulation for treatment of LBP or LDH has been practiced for hundreds of years. Theories for the effect of manipulation include restoring normal motion to restricted segments and impacts proprioceptive primary afferent neurons from paraspinal tissues. It also affects pain processing by altering the central facilitated state of the spinal cord.

Multiple randomized controlled trials and systematic review have been done to assess the efficacy of manual therapy. In a meta-analysis by Assendelft et al, spinal manipulation was found to be more effective than placebo for acute and chronic LBP.Santilli et al also found that active manipulation had more effect than simulated manipulation on pain relief of acute back pain and sciatica with disc protrusion. However, in a recent review article, the authors concluded that definitive values on safety and effectiveness of spinal manipulation cannot be made, but they admit that many patients with LDH did undergo manipulative treatment, and spinal manipulation may be effective in the treatment of symptomatic LDH.

The goal of surgery for a LDH is to remove the portion of disc that is impinging on the nerve root. There are many options for surgery for LDH, including open discectomy, laminotomy, laminectomy, or the combinations. There are also new techniques such as endoscopic discectomy, laser discectomy, and electrothermal disc decompression. Choice of surgery depends on surgeons' experience and condition of the patients. Favorable short-term results have been reported before.

Although lumbar traction, spinal manipulation, and surgery have been used extensively in the management of LDH, comparison of the three treatments has never been studied before. The purpose of this study is to compare the effect of lumbar traction, spinal manipulation, and surgery in the treatment of LDH.

ELIGIBILITY:
Inclusion Criteria:

* Age>20 and less than 80 y/o with LDH with moderate to severe (VAS pain > 4) LBP and/or sciatica. LDH should be proved by MRI of the lumbosacral spine. The duration of pain is less than 1 month.

Exclusion Criteria:

1. LBP probable due to serious spinal pathology such as spinal tumor, infection, and inflammatory disease such as ankylosing spondylitis.28
2. LDH with progressive weakness in the lower extremities or symptoms and signs suggesting cauda equina lesion.
3. Concomitant serious medical conditions.
4. History of spinal surgery before.
5. Severe osteoporosis or image studies suggesting instability of the lumbosacral spine.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
VAS pain score | Clinical evaluation will be conducted at pre-treatment, post-treatment day 7 and post-treatment 2 months after treatments.
  an 10-cm horizontal line will be used to assess average pain intensity in the last 1 week

SECONDARY OUTCOMES:
Global impression of change | Clinical evaluation will be conducted at pre-treatment, post-treatment day 7 and post-treatment 2 months after treatments.
  contains seven items from "very much improved" to "very much worse"
Modified Oswestry Disability Questionnaire (MODQ) | Clinical evaluation will be conducted at pre-treatment, post-treatment day 7 and post-treatment 2 months after treatments.
  For evaluation of disability related to LBP, Oswestry Disability Questionnaire (ODQ) is most widely used. ODQ is a 10-item self report instrument that evaluates perceived disability in 10 areas: pain intensity, ability to lift objects, ability to walk, ability to sit, ability to stand, ability to sleep, sex life, social life, traveling, and ability to complete personal hygiene activities. By using a 6-point Likert scale (0 = no limitation; 5 = severe limitation) , the total maximum scale is doubled and reported as a percentage of the patients perceived pain-related disability, with higher scores indicating greater disability. Because sex life could be an embarrassing issue in Chinese society, the investigators prefer to use modified or revised ODQ or MODQ,30,31 in which sex life is replaced by employment or homemaking. High validity and reliability of MODQ for LDH and LBP has been studied previously.
SF-36 | Clinical evaluation will be conducted at pre-treatment, post-treatment day 7 and post-treatment 2 months after treatments.
  The Medical Outcome Survey Short Form (SF-36) was used to assesses general health status. The SF-36 measures eight dimensions of health: general health perceptions, physical function, physical role, bodily pain, social functioning, mental health, emotional role, and vitality. The eight scales may be combined into two summary scores, the physical component summary (PCS) and the mental component summary (MCS). The SF-36 has well-established psychometric properties for the general population and individuals with LBP.

CONTACTS AND LOCATIONS:
Overall Officials: Lin-Fen Hsieh, M.D, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- ShinKongHospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided